CLINICAL TRIAL: NCT06634277
Title: Implementing a Patient Navigation Intervention Across a Health System to Address Treatment Entry Inequities
Brief Title: Philly NavSTAR Implementation Trial
Acronym: Philly NavSTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: Thomas Jefferson University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R61DA059033 (NIH); R61DA059033 (NIH)
Record Dates: First submitted 2024-02-03; First posted 2024-10-09 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Opioid Use Disorder
Keywords: patient navigation
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Single group pilot study with sequential implementation in 4 hospitals
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NavSTAR (Experimental): NavSTAR is a Patient Navigation service model to reduce internal and external barriers to recommended service engagement. It includes motivational interventions in tandem with proactive barrier resolution, targeting areas of addiction, medical, self-care, and basic needs.
  Interventions: Behavioral: NavSTAR (Philly adaptation)

INTERVENTIONS:
Behavioral: NavSTAR (Philly adaptation) — Patient Navigation

SUMMARY:
Patient Navigation (PN) interventions following hospitalization can reduce the differences that certain groups have been trying to access opioid use disorder treatment. These differences, which affect racial minority groups the most, contribute to the opioid overdose epidemic. However, delivering PN interventions on a wide scale requires many resources and coordination across institutions. This will use an evidence-based process to find solutions to these significant barriers by engaging community, hospital, and patient partners. This study is being conducted to learn more about how to implement NavSTAR, a patient navigation intervention for people with opioid use disorder, across a health system. Our research team showed in a previous study with 400 participants that NavSTAR significantly increased entry into opioid use disorder treatment, reduced readmissions to the hospital, and was highly cost- effective compared to treatment as usual. This study will first pilot NavSTAR with 32 patient participants across 4 hospitals in the City of Philadelphia. Then, we will conduct a large trial with 720 patient participants to see if we can reach people who need the intervention, and create a sustainable plan to continue the intervention after the grant award period.

DETAILED DESCRIPTION:
Opioid agonist treatment (OAT) is protective against overdose, yet less than 20% of people with opioid use disorder (OUD) engage in such treatment. Hospital utilization is high among people with OUD and can be a 'reachable moment' to initiate OAT. However, most hospitals lack the capacity to follow up with patients after discharge. Theory-based, empirically supported patient navigator (PN) interventions following hospital discharge reduce inequities in accessing community-based OAT by helping patients navigate complex systems of care. However, challenges persist in implementing PN interventions on a wide scale, as they require coordination across institutions, data sharing, dedicated personnel, and community resources. This is especially true in settings that reach diverse, resource-challenged communities. To bring these interventions to scale, strategies are needed to assess factors that influence PN implementation in hospitals to increase feasibility, reach, and sustainability. Testing innovative implementation strategies for PN interventions has the potential for significant impact, as it will demonstrate implementation success of an intervention that can address the opioid epidemic in real-world settings and close the research-to-practice translation gap. The proposed study is a type II hybrid implementation-effectiveness trial of Navigation Services To Avoid Rehospitalization (NavSTAR). Our research team showed in a single-site randomized trial with 400 participants that NavSTAR significantly increased OAT entry, reduced readmissions, and was highly cost-effective compared to treatment as usual. The present study will test an Implementation Facilitation (IF) strategy following Proctor's conceptual model using an external facilitator and an internal local clinical champion to provide training, resources, and performance feedback to implement NavSTAR in four hospitals. We hypothesize that engaging stakeholders (including patients, clinicians, and community leaders) in an IF strategy will create and test an implementation process that is feasible, acceptable, and effective in expanding access to OAT post-discharge. The R61 phase will conduct process mapping to identify existing hospital workflow and then refine an IF strategy through sequential pilot trials at 4 hospital sites in preparation for the R33 phase. The team's NavSTAR operations manual will be adapted to the sites to train the existing staff. R61 milestones include the creation of an implementation toolkit and data-sharing agreements.

The developmental R61 phase will focus on needs assessment and identifying IF strategies for system-wide adoption of NavSTAR in preparation for the R33 trial phase. This will be accomplished through four inter-related processes: 1) Process mapping with the CAB and CAP, 2) Conducting qualitative interviews to gain diverse stakeholder input, 3) Modifying the IF strategy, and 4) Conducting four short-duration, iterative pilot testing cycles in four hospitals to examine the IF strategy for feasibility and acceptability. Pilot testing will occur with existing personnel (master's level social workers) utilizing the NavSTAR manual of operations. Interviews with current participants in the pilot testing, organizational stakeholders, navigators, and clinician champions will be conducted both before and after the pilot testing cycles.

Aim 1: Providers, staff, organizational leadership, and patients at the four hospitals will be asked to participate in the study (N=40) by completing interviews about current navigation/ discharge processes and optimal IF strategies.

Aim 2: Patients will be recruited across four hospitals (8 at each hospital) to conduct a pilot trial (N=32) of NavSTAR implementation. The CAB/CAP feedback, stakeholder interviews, and results of the pilot testing cycles will inform the final implementation toolkit used in the R33 phase.

ELIGIBILITY:
Inclusion criteria:

1. age 18 or older;
2. current DSM-5 criteria for moderate to severe OUD;
3. willing and able to provide informed consent in English.

Exclusion criteria:

1. enrollment in OUD treatment 30-days prior to hospitalization;
2. residency outside the City of Philadelphia;
3. pregnancy;
4. planned discharge to a long-term inpatient care facility (e.g., hospice);
5. hospitalization for a suicide attempt.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-07-26 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Opioid Agonist Treatment (OAT) initiation | 3 months
  Post-discharge OAT initiation will be measured by self-report at follow-up, with verification through records where applicable (e.g., Community Behavioral Health system).

SECONDARY OUTCOMES:
Acceptability: Extent to which the intervention will be deemed acceptable by participants | 3 months
  Acceptability will be measured by the Acceptability of Intervention Measures Scale.
Appropriateness: Extent to which the intervention will be deemed appropriate by participants | 3 months
  Appropriateness will be measured using the Intervention Appropriateness Measure scale
Changes in Psychological distress from baseline to 3 months | Baseline to 3-month follow-up
  Kessler-6 Psychological Distress Scale (K6) will be used to assess how participants have been feeling (nervous, hopeless, restless, depressed, worthless, etc) during their last 30 days.
Opioid use (oral fluid) | 3 months
  Proportion of participants with positive oral fluid drug testing for opioids.
Changes in Social Support from Baseline to Follow-up | Baseline to 3 month follow-up
  Social support will be measured using the Social Support Scale to determine the extent to which services influenced social support.
Change in Recovery Capital from baseline to follow-up | Baseline to 3 month follow-up
  Recovery capital will be assessed using the BARC-10 scale.
Changes in Quality of Life from Baseline to Follow-up | Baseline to 3 month follow-up
  Quality of life will be measured via the WHOQOL-BREF instrument.
Self-reported days of opioid use in the past 30 days | Baseline to 3 month follow-up
  Self-reported days of non-medical opioid use in the past 30 days will be assessed at each interview.
Hospital Utilization | 3 months
  Information on acute care hospital utilization (including Emergency Department visits and Inpatient Admissions) will be assessed using health records and self-report (in the event of inconsistency, objective data will dominate).
Feasibility: Demonstrated ability to enroll participants in the intervention | From enrollment until end of follow-up (10 months)
  Feasibility will be measured by enrollment rate (Target 8 participants per month/per hospital), calculated as the number of eligible participants relative to the number screened. This is an implementation outcome measured in the aggregate (not patient-level)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Alexander, PhD, Principal Investigator — Friends Research Institute, Inc.; Jan Gryczynski, PhD, Principal Investigator — Friends Research Institute, Inc.
Locations (2):
- United States (2):
  - Jefferson Health, Philadelphia, Pennsylvania
  - Friends Research Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Because this is a feasibility pilot to inform a subsequent study, there is no plan to share IPD for the feasibility pilot. Interested researchers can nonetheless contact the PIs to discuss data sharing.

REFERENCES:
- [Background] Gryczynski J, Nordeck CD, Welsh C, Mitchell SG, O'Grady KE, Schwartz RP. Preventing Hospital Readmission for Patients With Comorbid Substance Use Disorder : A Randomized Trial. Ann Intern Med. 2021 Jul;174(7):899-909. doi: 10.7326/M20-5475. Epub 2021 Apr 6. PMID 33819055